CLINICAL TRIAL: NCT03937973
Title: The Effects of Social Experiences on Sleep and Cardiovascular Functioning
Brief Title: Social Experiences and Sleep Study
Acronym: SASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-24889; R01HL142051 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2019-05-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Sleep; Blood Pressure
Keywords: sleep; heart; stress

STUDY DESIGN:
Intervention Model Description: All participants will complete two nights in the sleep laboratory. One night will be a non-rejection control night. The other night will be a rejection task night. In this regard, African American and Caucasian American participants will be randomized to one of two conditions. All participants will be exposed to social rejection prior to bedtime; however, they will either be rejected by a person of their own race (in-group member) or a different race (out-group member)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blind to condition until the debriefing, which occurs the morning following the social-rejection task.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social rejection by in-group (Experimental): One hour prior to bed, participants will be exposed to a social rejection paradigm that includes a computerized ball-tossing game (Cyberball) and a speech task. Participants are made to believe that they are being rejected by someone of their own race/ethnicity (e.g., African American rejected by another African American).
  Interventions: Behavioral: Social rejection
- Social rejection by out-group (Experimental): One hour prior to bed, participants will be exposed to a social rejection paradigm that includes a computerized ball-tossing game (Cyberball) and a speech task. Participants are made to believe that they are being rejected by someone not of their own race/ethnicity (e.g., Caucasian American rejected by another African American).
  Interventions: Behavioral: Social rejection

INTERVENTIONS:
Behavioral: Social rejection — Social rejection paradigm

SUMMARY:
This study will test the effect of race-based social rejection on polysomnography derived sleep outcomes and nocturnal cardiovascular psychophysiology in a sample of 80 African Americans and 80 Caucasian Americans. The investigators will test group differences on these outcomes as well as within subjects by testing impact of rejection compared to a non-rejection control night in the sleep laboratory.

DETAILED DESCRIPTION:
African Americans (AA) are disproportionally burdened by cardiovascular disease compared to Caucasian Americans (CA). Poor sleep, which is more common among AA, may serve as an important pathway in understanding these disparities. Race-based rejection has been cross-sectionally related to poor sleep and negative cardiovascular outcomes. To test the links between social experiences and sleep, participants will spend two nights in the sleep laboratory. One night will be a control night where participants complete low arousal tasks prior to bedtime. On a second night, the investigators will randomize 80 AA and 80 CA to either race-based social rejection (i.e., being rejected by an out-group member) or same-race social rejection prior to bedtime to test the causal influences of race-based rejection on objective sleep parameters, measured using polysomnography, and nocturnal cardiovascular functioning. The investigators will test group differences on these outcomes as well as within subjects by testing impact of rejection compared to a non-rejection control night in the sleep laboratory. The order of the control and rejection task night will be counterbalanced.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 64 years old
* Self-identified as African American/Black or Caucasian American/White
* English speaking, able to provide consent
* Self-reported bedtime between 10PM and 12AM for 5/7 nights for the past 3 months (stability to be confirmed by sleep diary and wrist actigraphy).
* Self-reported sleep duration between 6.5 and 8.5 hours for 5/7 nights for the last month (duration to be confirmed by actigraphy and sleep diary)

Exclusion Criteria:

* Body mass index of 40 or above
* Participants at high risk for obstructive sleep apnea, based on "high risk" score from the STOP-Bang.
* Medical or psychiatric condition, as assessed by self-report and clinical interview that affect sleep and/or cardiovascular functioning, including doctor diagnosed arrhythmia, hypertension, congestive heart failure, major depression, bipolar disorder, post-traumatic stress disorder.
* Medication use that is likely to affect sleep and/or cardiovascular functioning, including antidepressants, anxiolytic or soporific medication, and beta-blockers.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in sleep onset latency, as determined by polysomnography | Assessed on the night of the social rejection task and compared to the control task night; it is anticipated that these nights will take place consecutively
  Sleep onset latency is the time (in minutes) from "lights out" to sleep onset on the nights following the social rejection task and the control task laboratory to onset of sleep, as measured via polysomnography

SECONDARY OUTCOMES:
Change in minutes of wake after sleep onset (WASO), as determined by polysomnography | Assessed on the night of the social rejection task and the night of the control task; it is anticipated that these nights will take place consecutively
  Number of minutes awake once sleep is initiated, measured via polysomnography on the nights following the social rejection task and the control task
Change in total sleep time, as determined by polysomnography | Assessed on the night of the social rejection task and the night of the control task; it is anticipated that these nights will take place consecutively
  Total number of minutes scored as sleep, measured via polysomnography on the nights following the social rejection task and the control task
Change in pre-ejection period (PEP) in response to rejection task | Baseline to Post-rejection task, anticipated average of 30 minutes
  Pre-ejection period is measured via impedance cardiography, averaged over a 5-minute baseline period and in the minutes during the rejection task
Change in heart rate variability (HRV) in response to rejection task | Baseline to Post-rejection task, anticipated average of 30 minutes
  Heart rate variability is measured via EKG, averaged over a 5-minute baseline period and in the minutes during the rejection task
Change in nocturnal heart rate variability | Assessed on the night of the social rejection task and the night of the control task; it is anticipated that these nights will take place consecutively
  Heart rate variability is measured via EKG, beginning at "lights out" and collected across the night following the rejection task and control task; it is anticipated that the two nights will occur consecutively.
Change in nocturnal pre-ejection period | Assessed on the night of the social rejection task and the night of the control task; it is anticipated that the two nights will occur consecutively
  Pre-ejection period will be measured by impedance cardiography, beginning at "lights out" and collected across the night following the rejection task and control task; it is anticipated that the two nights will occur consecutively.

CONTACTS AND LOCATIONS:
Overall Officials: Aric A Prather, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Our plan is to make all processed data available at the conclusion of the study in line with NIH guidelines
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All processed data should be available within 5 years of completion of the study
Access Criteria: Consistent with NIH guidelines